CLINICAL TRIAL: NCT06114433
Title: Development of 3D Printing High-Fidelity Upper Gastrointestinal Tract Model for Nursing Students in the Nasogastric Tube Training
Brief Title: Three-dimensional Upper Gastrointestinal Tract Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Group leader of Respiratory Therapists, Fu Jen Catholic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FJUH111192
Record Dates: First submitted 2023-10-28; First posted 2023-11-02 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Medical Education
Keywords: 3D printing; upper body manikin; upper gastrointestinal tract; nasogastric tube care; simulation-based training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional model group (Active Comparator): Received a regular learning
  Interventions: Other: Traditional model education
- 3D-printed presention group (Experimental): Received a regular learning plus 3D printing model
  Interventions: Other: 3D printed educational model

INTERVENTIONS:
Other: 3D printed educational model — Slide-based presention plus 3D printed educational model
  Arms: 3D-printed presention group
Other: Traditional model education — Slide-based presention plus traditional model
  Arms: Traditional model group

SUMMARY:
This study aims to develop an upper body manikin with a high-fidelity upper gastrointestinal tract and apply into the nasogastric tube training program for nursing students.

DETAILED DESCRIPTION:
Background：

Nursing trainees often fail to correctly prepare medical supplies and use stethoscopes for position assessment incorrectly when physicians perform nasogastric tube placement techniques. The traditional training model are expensive and difficult to access or maintain. It is easy to cause irreparable damage when repeated tearing and sticking of the elastic adhesive tape on the traditional model. Because of the high-priced the traditional model, it is impossible to use real milk, to simulate the nasogastric tube feeding. Inadequate clinical skills often raises patient safety concerns when assisting in changing nose pads and feeding. To enhance the nasogastric tube training for nursing students, the investigators used 3D-printed education model combined with clinical simulation-based training program.

Study Design：

This is a randomized controlled trial of medical education study.

Methods：

The investigators first designed our 3D upper body model using the 3D processing and analysis software. To create the basic outline of the 3D model, the investigators used a white-light handheld 3D scanner to scan a real human. To closely resemble the soft biological tissues of real human organs, an adequate material will be chosen in the study. The pre/post examination, student satisfaction, and direct observation of procedural skills will be used to evaluation the outcome of the study.

Effect：

The investigators expect the 3D-printed upper body manikin with a high-fidelity upper gastrointestinal tract model has potential in nasogastric tube training, particularly in helping trainees become familiar with the nasogastric tube care.

Keywords：

3D printing, upper body manikin, upper gastrointestinal tract, nasogastric tube care, simulation-based training

ELIGIBILITY:
Inclusion Criteria:

* Training at Fu Jen Catholic University Hospital.
* Signed the consent form.

Exclusion Criteria:

* Refused to participate in the study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Examination score of direct observation of procedural skills | immediately after the intervention
  maximun 100 and minimum 0, higher means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Yun Chao, PhD, Principal Investigator — Fu Jen Catholic University Hospital
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No